CLINICAL TRIAL: NCT04364165
Title: The Effect of Undetectable Equals Untransmittable (U=U) Messaging on HIV Testing Uptake Among South African Men: a Randomized Trial.
Brief Title: Effect of U=U Messaging on HIV in South Africa
Acronym: U=U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Desmond Tutu HIV Foundation (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 834483
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-07

CONDITIONS: HIV/AIDS
Keywords: Behavioral sciences; HIV testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care messaging (Experimental): On mobile clinic days randomized to standard of care messaging, participants will receive standard invitation cards distributed at the Tutu Tester containing basic information encouraging HIV testing. Messages will encourage men to come in for HIV testing at the mobile clinic on the same day. A mobile clinic recruiter will deliver the standard invitation card and share a brief script including the standard Tutu Tester message that free HIV testing is available at the Tutu Tester, with no further information or motivation to test.
  Interventions: Behavioral: Standard invitation to free HIV testing at mobile clinic
- U=U messaging (Experimental): On mobile clinic days randomized to U=U messaging, participants will receive the U=U invitation cards distributed at the Tutu Tester that will seek to assuage the fears of testing HIV positive by conveying the message that HIV treatment makes it possible for HIV positive people to be untransmittable and to live normal lives. Messages will encourage men to come in for HIV testing at the mobile clinic on the same day. A mobile clinic recruiter will deliver the U=U invitation card and share a brief script asking people if they knew they could control HIV and that pills exist that can keep them healthy and ensure they don't transmit the virus to their sex partners, and that free HIV testing is available at the Tutu Tester.
  Interventions: Behavioral: U=U messaging and invitation to free HIV testing at mobile clinic

INTERVENTIONS:
Behavioral: Standard invitation to free HIV testing at mobile clinic — Participants receive standard invitation to same day HIV testing at mobile clinic.
  Arms: Standard of care messaging
Behavioral: U=U messaging and invitation to free HIV testing at mobile clinic — Participants receive messaging about being undetectable equals untransmittable (U=U) and invitation to same day HIV testing at mobile clinic.
  Arms: U=U messaging

SUMMARY:
This cluster randomized trial will investigate whether messaging about being undetectable equals untransmittable (U=U) designed through a participatory, user-centered approach increases HIV testing uptake within men in Klipfontein Mitchells Plain (KMP) district in Cape Town, South Africa.

DETAILED DESCRIPTION:
This study will investigate the effect of participatory, user designed messaging to increase knowledge about U=U on HIV testing uptake within men in the Klipfontein Mitchells Plain (KMP) district, a resource-limited, densely populated, high HIV disease burden area in Cape Town, through a cluster randomized trial design. The study will be conducted in two phases: Phase 1 is a participatory, human-centered design framework will be used to develop U=U messages to increase HIV testing uptake in men. Phase 2 is a cluster randomized trial that will determine the effect of U=U messaging on HIV testing uptake. The primary outcome will be HIV testing uptake at a community-based mobile clinic. Secondary outcomes will include the proportion of males tested who are HIV-positive (and newly HIV positive).

Men in the intervention group will receive invitation cards for mobile HIV testing that contain U=U messages. Men in the control group will receive invitation cards for mobile HIV testing that contain standard messaging. Mobile clinic days (i.e. clusters of men receiving invitation cards on a single day) will be the unit of randomization. Recruitment will be conducted by trained mobile clinic staff at high foot-traffic sites in the KMP community. Recruitment efforts will be focus on young men in multiple mobile testing sites that are located in areas within KMP.

ELIGIBILITY:
Inclusion Criteria:

* Men at least 18 years of age within the vicinity of the mobile Tutu Tester HIV testing mobile clinic

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1048 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Buttenheim, PhD, Principal Investigator — University of Pennsylvania; Dvora Joseph Davey, Principal Investigator — Desmond Tutu HIV Foundation
Locations (1):
- Desmond Tutu HIV Foundation, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Smith PJ, Joseph Davey DL, Schmucker L, Bruns C, Bekker LG, Medina-Marino A, Thirumurthy H, Buttenheim AM. Participatory Prototyping of a Tailored Undetectable Equals Untransmittable Message to Increase HIV Testing Among Men in Western Cape, South Africa. AIDS Patient Care STDS. 2021 Nov;35(11):428-434. doi: 10.1089/apc.2021.0101. PMID 34739334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Peer promoters were trained to deliver brief messages to men at selected high foot-traffic sites in the KMP community. Males ≥ 18 years of age within the vicinity of the mobile Tutu Tester HIV testing van and willing to consent to participate in the study were eligible for inclusion.
Units Other Than Participants: Mobile clinic days
Period: Overall Study
Arm/Group | Standard of Care Messaging | U=U Messaging
Started | 544; 20 Mobile clinic days | 504; 20 Mobile clinic days
Completed | 68; 5 Mobile clinic days | 112; 7 Mobile clinic days
Not Completed | 476; 15 Mobile clinic days | 392; 13 Mobile clinic days

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Messaging: Participants randomized into this arm will receive standard invitation cards distributed at the Tutu Tester containing basic information encouraging HIV testing. Messages will encourage men to come in for HIV testing at the mobile clinic on the same day. A mobile clinic recruiter will deliver the standard invitation card and share a brief script including the standard Tutu Tester message that free HIV testing is available at the Tutu Tester, with no further information or motivation to test.
  Standard invitation to free HIV testing at mobile clinic: Participants receive standard invitation to same day HIV testing at mobile clinic.
- U=U Messaging: Participants randomized into this arm will receive the U=U invitation cards distributed at the Tutu Tester that will seek to assuage the fears of testing HIV positive by conveying the message that HIV treatment makes it possible for HIV positive people to be untransmittable and to live normal lives. Messages will encourage men to come in for HIV testing at the mobile clinic on the same day. A mobile clinic recruiter will deliver the U=U invitation card and share a brief script asking people if they knew they could control HIV and that pills exist that can keep them healthy and ensure they don't transmit the virus to their sex partners, and that free HIV testing is available at the Tutu Tester.
  U=U messaging and invitation to free HIV testing at mobile clinic: Participants receive messaging about being undetectable equals untransmittable (U=U) and invitation to same day HIV testing at mobile clinic.
- Total: Total of all reporting groups
Arm/Group | Standard of Care Messaging | U=U Messaging | Total
Number analyzed (Participants) | 68 | 112 | 180
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [26 to 44] | 35 [28 to 46] | 35 [27 to 45]
Sex: Female, Male [Count of Participants; unit: Participants] — Only men were eligible for recruitment into the study.
  Participants
    Female | 0 | 0 | 0
    Male | 68 | 112 | 180
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or mixed race | 68 | 112 | 180
Region of Enrollment [Number; unit: participants] — Recruitment took place in the Klipfontein Mitchells Plain (KMP) District in Cape Town, Western Cape Province, South Africa.
  participants
    South Africa | 68 | 112 | 180

OUTCOME MEASURES:

1. Primary Outcome: HIV Testing Uptake
Description: Number of Participants that were Invited and Came for HIV Testing
Time Frame: Recruitment took place over 12 days.
Population: The unit of randomization was Mobile Clinic Days; analysis of outcome measures summarizes the individual Number of Participants, or number of men who received the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Messaging | U=U Messaging
Number analyzed (Participants) | 544 | 504
Participants | 68 | 112
Statistical Analysis 1: Comparison: Standard of Care Messaging vs U=U Messaging; Test type: Superiority; p = .01, Regression, Logistic; Odds Ratio (OR) = 2, 95% CI 2-sided [1.44 to 2.78]

2. Secondary Outcome: HIV Positivity
Description: Number of Participants that Came for Testing and Obtained an HIV-Positive Result
Time Frame: Recruitment took place over 12 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Messaging | U=U Messaging
Number analyzed (Participants) | 68 | 112
Participants | 3 | 7
Statistical Analysis 1: Comparison: Standard of Care Messaging vs U=U Messaging; Test type: Superiority; p = .41, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.36 to 5.78]

ADVERSE EVENTS:
Time Frame: 1 day from recruitment
Arm/Group | Standard of Care Messaging | U=U Messaging
All-Cause Mortality (participants affected / at risk) | 0/544 | 0/504
Serious Adverse Events (participants affected / at risk) | 0/544 | 0/504
Other Adverse Events (participants affected / at risk) | 0/544 | 0/504

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT04364165/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT04364165/ICF_001.pdf